CLINICAL TRIAL: NCT05193903
Title: Evaluation of an Interactive Risk Information Tool to Increase COVID-19 Vaccination Incidence in Vaccine-hesitant People During Omicron Wave in Germany
Brief Title: Evaluation of an Interactive Risk Information Tool to Increase COVID-19 Vaccination Incidence in Vaccine-hesitant People
Acronym: iWILL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Medical Center Mainz (Other); Max Planck Institute for Human Development (Other); Federal Joint Committee (Other Government)
Responsible Party: Principal Investigator, Odette Wegwarth, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VSF1_2021-194
Record Dates: First submitted 2021-12-14; First posted 2022-01-18 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Infection
Keywords: COVID-19 vaccination, vaccine-hesitancy
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Intervention Model Description: 1 intervention group, 1 control group (Cross-sectional study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Simulation (Experimental): Interactive information tools
  Interventions: Behavioral: Simulation
- Control: Text (Other): Standard text-based information
  Interventions: Behavioral: Text

INTERVENTIONS:
Behavioral: Simulation — The participants in the intervention group receive two interactive simulations in addition to a general text module that provides sequential, animated information on the spread of the virus without prevention, the effectiveness of vaccination and potential side effects of vaccination on a herd protection level and the individual level.
  Arms: Intervention: Simulation
Behavioral: Text — The participants in the control group receive two text-based information in addition to a general text module that provides information on the spread of the virus without prevention, the effectiveness of vaccination and potential side effects of vaccination on a herd protection level and the individual level.
  Both conditions ensure the provision of a level of knowledge that at least corresponds to standard care.
  Arms: Control: Text

SUMMARY:
Coronavirus (COVID-19) vaccines have saved millions of lives since release and remain a key tool in the fight against the pandemic.

However, most countries have not reached the vaccine uptake rates needed to relieve pressure on hospitals and intensive care units (ICUs) during peak corona periods. Reduced effectiveness of vaccines in preventing infections with the Omicron variant and milder courses of the disease may trigger and support beliefs that vaccination is no longer necessary, especially among vaccine sceptics.The term 'vaccine sceptic', however, is used heterogeneously and often interchangeably to describe both 'vaccine hesitants' and 'vaccine deniers'. In contrast to vaccine deniers, characterized by a definite and unwavering decision not to get vaccinated, vaccine hesitants are characterized by a spectrum of indecisiveness, with a high need for information on both benefits and harms. They may still decide to get vaccinated if information succeeds in convincing them. In light of the potential for a change of mind in vaccine-hesitants the key question is: How does one best address their high needs for balanced risk ratio information? Evidence from cognitive and behavioral science suggests that interactive simulations of risk information, which imitate mechanisms by which humans sequentially and experientially sample risk information naturally, can be more effective in helping people develop adequate risk perceptions and initiate behavioral change than the ubiquitously used conventional text-based formats. The study therefore seeks to determine if interactive risk ratio simulation relative to a text-based format are more effective in prompting positive change in unvaccinated, vaccine-hesitant respondents' intention to get the COVID-19 and also in the respective benefit-to-harm ratio assessment during the Omicron wave in Germany.

DETAILED DESCRIPTION:
The iWILL study is a cross sectional study that aims to evaluate the effectiveness of interactive risk ratio simulation (intervention) relative to a text-based format (control) in COVID-19 vaccine-hesitant people in Germany.

The objectives of iWILL are:

1. to adapt the already piloted, digital, interactive, evidence-based counseling tool ExploreVac (focus on herd protection) as well as a new simulation (focus on individual protection) to the most current evidence (including age adjustment) for communicating vaccine effectiveness and side effects as evidence-based patient information using the example of COVID-19 vaccination,
2. to implement the adapted version of ExploreVac and the new simulation in care with the aim to increase the vaccination incidence among vaccine hesitant individuals, to improve their subjective assessment of vaccination's benefits and harms, and to reduce the presumed increased counseling effort of the GP compared to standard care,
3. to test whether the intervention is superior as compared to the control on these endpoints,
4. to draw conclusions about the transferability of the developed method for other established vaccinations (HPV, influenza protection) and vaccinations for future infectious diseases.

Primary hypothesis:

(H1) The intervention group (interactive simulations) will show a higher positive change (T0/baseline to T1/after intervention) in vaccination intention than the control group (text-based information).

Secondary hypotheses:

(H2) The intervention group (interactive simulations) will show a higher positive change (T0/baseline to T1/after intervention) in their positive subjective benefit-to-harm assessment of the COVID-19 vaccine's benefit-to-harm ratio than does the control group.

(H3) The intervention group reports a lower need for additional counseling by their GPs than does the control group.

(H4) The intervention group (interactive simulations) will show a higher correspondence between their intended behavior (T1) and their actual reported vacccinataion behavior (T2/ follow-up after 6 months).

Recruitment of unvaccinated, vaccine hesitant German residents will be established by using probability-based internet panels maintained by respondi (Cologne, Germany). The study will be pursued with cross-sectional national sample.

Intervention condition: two interactive simulations informing 1) about absolute risks of infection, hospitalization, ICU admission, and death after exposure to COVID-19 relative to vaccination's side effects (e.g., myocarditis in men ≤35 years) in 100,000 vaccinated and 100,000 unvaccinated individuals, all adjustable to four different age groups (18- 34 years, 35-59 years, 60-79 years, ≥ 80 years due to considerable differences in each of the depicted risks (Supplement) and 2) about the benefits of vaccination for the population as a whole (herd) in terms of preventing infections and deaths.

Control condition (see also below): two text module informing 1) about absolute risks of infection, hospitalization, ICU admission, and death after exposure to COVID-19 relative to vaccination's side effects (e.g., myocarditis in men ≤35 years) in 100,000 vaccinated and 100,000 unvaccinated individuals, all adjustable to four different age groups (18- 34 years, 35-59 years, 60-79 years, ≥ 80 years due to considerable differences in each of the depicted risks (Supplement) and 2) about the benefits of vaccination for the population as a whole (herd) in terms of preventing infections and deaths.

The educative information material in both conditions is based on non-directive evidence-based patient counseling according to the guideline on evidence-based health information. After the study condition, participants are informed that any further questions about vaccination can be discussed with the GP.

The questionnaire at T0 (baseline) and T1 (directly after the intervention) takes maximum 10 minutes to complete (without exploration of intervention material). Given that participants are free to spend as much time as participants want with the educative information material, the total survey time can be longer, however.

About six months after first participation in the study, participants are re-contacted via e-mail and are asked to fill out a second questionnaire (6-months follow-up, T2), which approximately takes about 5 minutes to complete to learn more about potential the translation of the intention into vaccination behavior.

ELIGIBILITY:
Inclusion Criteria:

* Hesitancy towards COVID-19 vaccination
* Not yet vaccinated against COVID-19
* Age ≥ 18 years.

Exclusion Criteria:

* No hesitancy towards COVID-19 vaccination
* Already vaccinated
* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1188 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline vaccination intention at T1 | Immediately after Intervention (T1)
  Change in 5-point response scale of vaccination intention between baseline and post-intervention judgement "I will definitely get the COVID-19 vaccination"; "I will probably get the COVID-19 vaccination"; "I am unsure if I will get the COVID-19 vaccination"; "I will probably not get the COVID-19 vaccination", and "I will definitely not get the COVID-19 vaccination."
  NOTE: This scale is categorical, that means values are only used to distinguish between the 5 categories and DO NOT indicate better or worse outcomes.

SECONDARY OUTCOMES:
Change from baseline assessment of vaccine-related benefiit-to-harm at T1 | Immediately after Intervention (T1)
  Change in 5-point response scale of vaccine-related benefiit-to-harm assessment
  The beneﬁts of the COVID-19 vaccination clearly outweigh the harms," "The beneﬁts of the COVID-19 vaccination somewhat outweigh the harms," "Beneﬁts and harms of the COVID-19 vaccination are balanced," "The harms of the COVID-19 vaccination somewhat outweigh the beneﬁts," "The harms of the COVID-19 vaccination clearly outweigh the beneﬁts."
  NOTE: This scale is categorical, that means values are only used to distinguish between the 5 categories and DO NOT indicate better or worse outcomes.
Number of GP counselings at 6-months follow-up | 6-months follow up (T2)
  Measured by the number of visits of the GP to receive additional counselling on the vaccine after study intervention/control
Actual vaccination behavior at T2 | 6-months follow up (T2)
  Used to check for correspondence between vaccination intention expressed at T1 and actual behvavior at T2

CONTACTS AND LOCATIONS:
Overall Officials: Odette Wegwarth, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided